CLINICAL TRIAL: NCT06620614
Title: Comparative Study on Fractionated Versus Bolus Dose of Hyperbaric Bupivacaine in Patients Undergoing Transurethral Resection of Prostate Surgery Under Subarachnoid Block.
Brief Title: A 3 Months Duration Interventional Study Comparing Hemodynamic Parameters Between Bolus and Fractionated Group.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Academy of Medical Sciences, Nepal (Other Government)
Responsible Party: Principal Investigator, Shushma K C, Doctor, National Academy of Medical Sciences, Nepal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 187/2079/80
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Prostatic Hyperplasia, Benign
Keywords: Fractionated Dose; Heavy Bupivacaine; Spinal Anesthesia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: An approval from the Institutional Review Board (IRB), NAMS was taken prior to commencing the study. 72 Patients of ASA physical status I or II scheduled for Transurethral Resection of prostate under Sub-arachnoid block were enrolled in the study. . Patient's characteristics including name, gender, age, body weight, height and body mass index were recorded.
  Patients were kept nil per oral as per American society of anesthesiologist guidelines prior to surgery. Study pouplation were divided into two groups:
  * Bolus group
  * Fractionated group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fractionated group arm (Experimental): In this group ,participants are given 1.6 ml of Injection Heavy Bupivacaine 0.5% initially followed by 0.9ml after 60 seconds at a rate of 0.2ml/hr.
  Interventions: Combination Product: 0.5% Heavy Bupivacaine
- Bolus arm group (Placebo Comparator): In this group ,participants are given Injection Heavy Bupivacaine 0.5% 2.5ml bolus at a rate of 0.2ml/hr
  Interventions: Combination Product: 0.5% Heavy Bupivacaine

INTERVENTIONS:
Combination Product: 0.5% Heavy Bupivacaine — There are two groups.
  Other Names: 26 G Quincke's needle

SUMMARY:
The goal of this study is to compare the intraoperative hemodynamic status, characteristics of block of fractionated versus single bolus dose of Hyperbaric Bupivacaine in patient undergoing Transurethral Resection of Prostate(TURP) surgery under Subarachnoid block(SAB).

Seventy-two patients aged 50 years and above belonging to American Physical status I and II are divided into two study group.

Group B will receive Injection 0.5 % hyperbaric bupivacaine 2.5 ml single bolus dose and group F will receive same concentration and volume of hyperbaric bupivacaine with two third dose initially (i.e. 1.6 ml) and remaining one third dose (i.e. 0.9 ml) after 60 seconds at the rate of 0.2ml/sec.

DETAILED DESCRIPTION:
The aim of this study is to compare the intraoperative hemodynamic status, characteristics of block of fractionated versus single bolus dose of Hyperbaric Bupivacaine in patient undergoing TURP surgery under SAB.

Seventy-two patients aged 50 years and above belonging to American Physical status I and II undergoing transurethral resection of prostate for benign enlargement of prostate under subarachnoid block are enrolled and are divided into two groups having 36 patients in each.

Group B will receive Injection 0.5 % hyperbaric bupivacaine 2.5 ml single bolus dose and group F will receive same concentration and volume of hyperbaric bupivacaine with two third dose initially (i.e. 1.6 ml) and remaining one third dose (i.e. 0.9 ml) after 60 seconds at the rate of 0.2ml/sec.

Intraoperative mean arterial pressure (MAP), heart rate, onset of sensory and motor block, duration of sensory and motor block, and total intraoperative consumption of vasopressor are observed and compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50 years and above patients undergoing TURP surgery under SAB
* American Society of Anesthesiologist's Physical Status: I and II.

Exclusion Criteria:

* Patients with history of uncontrolled hypertension.
* Patients with previous history of cerebrovascular accidents.
* Patients with history of spinal deformity.
* Patients with known allergy to local anesthetics.
* Patient with Infection at site of injection.
* Patient with history of coagulopathy.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All male participants from 50 years and above
Enrollment: 72 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Comparision of mean arterial pressure(MAP) in both participants with subarachnoid block | Throughout study completion,an average of 3 months
  Hypotension was defined when mean arterial pressure (MAP) decreased ≤20% from baseline.
Comparision of heart rate in both participants with subarachnoid block | Throughout study completion,an average of 3 months
  Bradycardia was defined when heart rate is less than 60 beats per minute.
Comparision of total consumption of vasopressors used during intraoperative period between the groups. | Throughout study completion,an average of 3 months
  Injection Mephentermine 6mg iv was given for hypotension

SECONDARY OUTCOMES:
Comparision of time for onset of sensory between the groups. | Throughout study completion,an average of 3 months.
  Sensory block was assessed by loss of sensation to pinprick with blunted tip needle bilaterally in the dermatomal levels. It was tested every 3 min until achievement of maximum sensory block i.e. till T10 level
Comparision of time for onset of motor block between the groups | Throughout study completion,an average of 3 months.
  Time required to reach Modified Bromage scale =3, where Bromage 0= no motor block ,Bromage 3= complete block of motor limb
Comparision of the time of regression of sensory block between two groups. | Throughout study completion,an average of 3 months
  Loss of pinprick sensation every 30 minutes postoperatively until it reached the S2 segment
Comparision of the time of regression motor block between two groups. | Throughout study completion,an average of 3 months.
  Assessed every 30 minutes postoperatively Time required to reach Modified Bromage scale =0, where Bromage 0= no motor block ,Bromage 3= complete block of motor limb.
Comparision of adverse effects like nausea, vomiting and shivering between the groups | Throughout study completion,an average of 3 months.
  Side effects managed according to hospital protocol

CONTACTS AND LOCATIONS:
Overall Officials: Pusparaj Poudel, MD, Study Chair — Bir Hospital
Locations (1):
- National Academy of Medical Sciences, Bir Hospital, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nash J. Benign prostatic hyperplasia: prevalence and diagnosis. GM Journal. 2010;40:321-4
- [Background] Persu C, Georgescu D, Arabagiu I, Cauni V, Moldoveanu C, Geavlete P. TURP for BPH. How large is too large? J Med Life. 2010 Oct-Dec;3(4):376-80. PMID 21254734
- [Background] Bhattacharyya S, Bisai S, Biswas H, Tiwary MK, Mallik S, Saha SM. Regional anesthesia in transurethral resection of prostate (TURP) surgery: A comparative study between saddle block and subarachnoid block. Saudi J Anaesth. 2015 Jul-Sep;9(3):268-71. doi: 10.4103/1658-354X.158497. PMID 26240544
- [Background] Gandhi M, Kabir KK, Arora KK, Tiwari K. Comparative study between fractionated and single bolus dose of local anaesthetic in elective lower segment caeserean section. Indian J Clin Anaesth. 2019;6(3):386-90
- [Background] Kararmaz A, Kaya S, Turhanoglu S, Ozyilmaz MA. Low-dose bupivacaine-fentanyl spinal anaesthesia for transurethral prostatectomy. Anaesthesia. 2003 Jun;58(6):526-30. doi: 10.1046/j.1365-2044.2003.03153.x. PMID 12846615
- [Background] Beed M. Anaesthesia for gynaecological and genitourinary surgery. In: Aitkenhead A, Thompson J, Rowbotham D, Moppett I, editors. Smith and Aitkenhead's Textbook of Anaesthesia. 6 th edition. London: Churchill Livingstone/Elsevier; 2013. p. 568-77
- [Background] Puri N, Talwar A. Comparative Study of Ephedrine and Mephertermine in Treatment of Hypotension in Patients Undergoing Elective Trans Urethral Resection Prostate (TURP). Journal of Bangladesh College of Physicians and Surgeons. 2010;28(1):10-6
- [Background] Favarel-Garrigues JF, Sztark F, Petitjean ME, Thicoipe M, Lassie P, Dabadie P. Hemodynamic effects of spinal anesthesia in the elderly: single dose versus titration through a catheter. Anesth Analg. 1996 Feb;82(2):312-6. doi: 10.1097/00000539-199602000-00017. PMID 8561333
- [Background] Nugroho AM, Sugiarto A, Chandra S, Lembahmanah L, Septica RI, Yuneva A. A Comparative Study of Fractionated Versus Single Dose Injection for Spinal Anesthesia During Cesarean Section in Patients with Pregnancy-Induced Hypertension. Anesth Pain Med. 2019 Feb 6;9(1):e85115. doi: 10.5812/aapm-85115. eCollection 2019 Feb. PMID 30881909
- [Background] Norris MC. Neuraxial anaesthesia. In: Barash PG, Cullen BF, Stoelting RK, Cahalan MK, Stock MC, Ortega R, Sharar SM, Holt NF, editors. Clinical Anaesthesia. 8 thedition. New Delhi: Wolters Kluwer; 2017. p. 914-44.
- [Background] Brull R, Macfarlane AJ, Chan VW. Spinal, epidural, and caudal anaesthesia. In: Miller RD, editor. Miller's anaesthesia. 8 th edition. Philadelphia: Elsevier Saunders;2015. p. 1684-720.
- [Background] Badheka JP, Oza VP, Vyas A, Baria D, Nehra P, Babu T. Comparison of fractionated dose versus bolus dose injection in spinal anaesthesia for patients undergoing elective caesarean section: A randomised, double-blind study. Indian J Anaesth. 2017 Jan;61(1):55-60. doi: 10.4103/0019-5049.198390. PMID 28216705
- [Background] Ramasali M.V., Vankaylapatti S. D., Appagalla S, Kulkarni D. K., Pasupuleti S. A Prospective Randomised Double-Blind Comparative Study of Bolus versus Fractionated Dose Injection in Spinal Anaesthesia for Pregnant Women undergoing elective Caesarean Section. Indian J Anesth Anal 2018; 5(11):1840-45
- [Background] Derakhshan P, Faiz SHR, Rahimzadeh P, Salehi R, Khaef G. A Comparison of the Effect of Fractionated and Bolus Dose Injection on Spinal Anesthesia for Lower Limb Surgery: A Randomized Clinical Trial. Anesth Pain Med. 2020 Aug 23;10(5):e102228. doi: 10.5812/aapm.102228. eCollection 2020 Oct. PMID 34150559
- [Background] Kaniyil S, Priya PG, Nithinkumar MP, Sneha SR. Fractional spinal anaesthesia in high-risk elderly patients for orthopaedic surgery - Case series. Indian J Anaesth. 2023 Jul;67(7):651-654. doi: 10.4103/ija.ija_888_22. Epub 2023 Jul 14. PMID 37601939
- [Background] Tiwari K, Masar R. Comparison Between Fractionated and Single Bolus Dose of Local Anaesthetic (Bupivacaine 0.5% Heavy) in Elective Lower Segment Caeserean Section. Int. J. Health Clin. Res. 2020; 3(6):36-42
- [Background] Srivastava N, Ahluwalia P, Jheetay GS, Singh G. Bolus dose versus fractionated dose injection of hyperbaric bupivacaine in spinal anaesthesia among adult patients undergoing lower limb surgery: A prospective study. Indian J Clin Anaesth. 2020;7(2):238-44
- [Background] Hossain MM, Biswas B, Mohanta PK, Hassan MM, Basu P, Islam F. Comparison between fractionated dose with bolus dose in Spinal Anaesthesia for haemodynamic stability and duration of analgesia in patients undergoing elective Lower Segment Caesarean Section (LSCS). Mediscope. 2020 Sep 29;7(2):95-102
- [Background] Sowmya NL. Comparison of Fractionated versus Bolus Dose Injection of Drug in Spinal Anaesthesia for Lower Limb Surgeries. Int. J. Sci. Res. 2020;Vol 9
- [Background] Mahbuba S, Chy MM, Naz S, Begum M, Jahan SS, Sheikh ZA. Comparison of sensory and motor block outcome of fractionated versus single bolus dose administration of hyperbaric bupivacaine in elective cesarean section. Medico Research Chronicles. 2021 ;8(4):317-24
- See also: This study describes about prevalence of benign prostatic hyperlasia in elderly male. — https://pavilionhealthtoday.com/gm/benign-prostatic-hyperplasia-prevalence-and-diagnosis/
- See also: This article describes about TURP for Benign Prostatic Hyperplasia — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3019067/
- See also: This article describes about comparision between saddle and subarachnoid block in TURP surgery. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4478818/
- See also: This article describes about Low-dose bupivacaine-fentanyl spinal anaesthesia for transurethral prostatectomy. — https://pubmed.ncbi.nlm.nih.gov/12846615/
- See also: This is academic book of anesthesia — https://books.google.com.np/books/about/Smith_and_Aitkenhead_s_Textbook_of_Anaes.html?id=VZBSAAAAQBAJ&redir_esc=y
- See also: This study describes about comparison of Ephedrine and Mephertermine in Treatment of Hypotension in Patients Undergoing Elective Trans Urethral Resection Prostate (TURP). — https://www.banglajol.info/index.php/JBCPS/article/view/4638
- See also: This study describes about Hemodynamic effects of spinal anesthesia in the elderly: single dose versus titration through a catheter. — https://pubmed.ncbi.nlm.nih.gov/8561333/
- See also: This study describes about comparision of fractionated versus single dose injection for spinal anesthesia during cesarean section in patients with pregnancy-induced hypertension — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6413406/
- See also: This is academic book of anesthesia — https://anesthesiology.lwwhealthlibrary.com/book.aspx?bookid=2137
- See also: This is academic book of anesthesia — https://www.dr-mustafazakaria.org/miller_s-basics-of-anesthesia-2023-8th-edition/
- See also: This study compares between fractionated dose versus bolus dose injection in spinal anaesthesia for patients undergoing elective caesarean section: — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5296809/
- See also: This study compares between Fractionated and Bolus Dose Injection on Spinal Anesthesia for Lower Limb Surgery — https://pubmed.ncbi.nlm.nih.gov/34150559/
- See also: This study compares between Fractional spinal anaesthesia in high-risk elderly patients for orthopaedic surgery — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10436721/
- See also: This study compares between Fractionated and Single Bolus Dose of Local Anaesthetic (Bupivacaine 0.5% Heavy) in Elective Lower Segment Caeserean Section — https://core.ac.uk/download/pdf/335018765.pdf
- See also: This study compares between fractionated dose with bolus dose in Spinal Anaesthesia for haemodynamic stability and duration of analgesia in patients undergoing elective Lower Segment Caesarean Section — https://pdfs.semanticscholar.org/b3c5/beacd5a02cc5619d71b2774a16a01d0399fa.pdf
- See also: This study compares between Fractionated versus Bolus Dose Injection of Drug in Spinal Anaesthesia for Lower Limb Surgeries — https://www.ijsr.net/archive/v9i1/ART20204456.pdf
- See also: This study compares between sensory and motor block outcome of fractionated versus single bolus dose administration of hyperbaric bupivacaine in elective cesarean section — https://medrech.com/index.php/medrech/article/view/520